CLINICAL TRIAL: NCT01179152
Title: Childhood Asthma and Return to School: the September Epidemic Exacerbation in Israel.A Controlled Trial of the Effectiveness of Preventive Treatment With Symbicort or Budicort Turbuhaler
Brief Title: Study of Preventive Treatment With Symbicort or Budicort Turbohaler in Childhood Asthma Return to School Epidemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hermanasthma
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Asthma Exacerbation
Keywords: asthma, september epidemic, children, preventive
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Budicort (Active Comparator): 75 children will receive treatment with Budicort 200 mcg
  Interventions: Drug: Budesonide turbuhaler, Budesonide+Formoterol turbuhaler
- Symbicort (Active Comparator): 75 children will receive treatment with Symbicort 160 mcg
  Interventions: Drug: Budesonide turbuhaler, Budesonide+Formoterol turbuhaler
- counselling (No Intervention): 75 children who will not treated as their request but will be folowedup
  Interventions: Drug: Budesonide turbuhaler, Budesonide+Formoterol turbuhaler

INTERVENTIONS:
Drug: Budesonide turbuhaler, Budesonide+Formoterol turbuhaler — Budesonide 200 mcg turbuhaler or Budesonide+Formoterol 160mcg turbuhaler
  Other Names: Budesonide turbuhaler; Budesonide+Formoterol turbuhaler

SUMMARY:
During the second week of September( week 38 of the year)there are recorded data of exacerbation of asthma all over the world, including Israel. A short preventive treatment of 6 weeks may reduce asthma exacerbation in children,reduce primary care and ER visiting and hospitalization.

DETAILED DESCRIPTION:
During the second week of September( week 38 of the year)there are recorded data of exacerbation of asthma all over the world, including Israel. A short preventive treatment of 6 weeks may reduce asthma exacerbation in children,reduce primary care and ER visiting and hospitalization.

We will study the effectiveness of Budicort or Symbicort turbuhaler as a preventive treatment in children aged 6-18 years.

ELIGIBILITY:
Inclusion Criteria:

age : 6-18 years suffering from asthma asthma exacerbation during 1/9/2009-15/10/2009

-

Exclusion Criteria:

any chronic condition that can involve respiratory tract (other than asthma) treated as prevention with ICS or montelukast from July 2010 Treated with oral steroids during the August 2010 asthma exacerbation one week prior study inclusion

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
reduction of asthma exacerbation during the study period | An average time of 8 weeks
  less asthma exacerbation

SECONDARY OUTCOMES:
less primary care physician visits | An average time of 8 weeks
  less primary care physician visits less ER visits less hospitalization due to asthma exacerbation

CONTACTS AND LOCATIONS:
Overall Officials: Avner He Cohen, Dr, Principal Investigator — Clalit Health Services
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- [Background] Johnston NJ, Johnston SL, Duncan JM, Greene JM,Keith PK,Roy M, Wsaerman S, Sears MR. The september epidemic of asthma exacerbation in children:a search for etiology. J allergy Clin Immunol 2005,115;132-8 Scheuerman O, Meyerowitch J, Marcus N, Hoffer V, Batt E , Garty B-Z. The september epidemic of asthma in Israel. J of Asthma 2009;46;652-5 Johnston NW, Mandhane PJ, Dai J, Duncan JM, Greene JM,Lambert K, Sears Mr. Attenuation of the september epidemic of asthma exacerbation in children: A randomized controlled trial of montelukast added to usual therapy. Pediatrics;120;e702-e712.